CLINICAL TRIAL: NCT01740505
Title: HealthySteps: A Pilot Randomized Controlled Trial of Exercise to Improve Walking Energetics, Fatigue, and Activity in Older Adults With Mobility Limitation
Brief Title: HealthySteps: Exercise for Older Adults With Mobility Limitation
Acronym: HealthySteps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Drummond Foundation (Unknown)
Responsible Party: Principal Investigator, Dawn C. Mackey, Assistant Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFMG-001
Record Dates: First submitted 2012-11-23; First posted 2012-12-04 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Mobility Limitation
Keywords: energy cost of walking; energy metabolism; aged; older adult; exercise; gait; walking; aerobic; motor skill
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Timing and Coordination (Experimental)
  Interventions: Behavioral: Timing and Coordination
- Aerobic Walking (Experimental)
  Interventions: Behavioral: Aerobic Walking
- Stretching and Relaxation (Active Comparator)
  Interventions: Behavioral: Stretching and Relaxation

INTERVENTIONS:
Behavioral: Timing and Coordination — This intervention is based on progressively difficult stepping and walking patterns that promote the timing and coordination of stepping within the gait cycle. Small-group 60-minute classes twice weekly for 12 weeks.
  Arms: Timing and Coordination
Behavioral: Aerobic Walking — Outdoor walking with progressive increases in exercise intensity. Small-group 60-minute classes twice weekly for 12 weeks.
  Arms: Aerobic Walking
Behavioral: Stretching and Relaxation — Full-body stretching, range-of-motion exercises, and relaxation techniques. No specific gait training. Small-group 60-minute classes twice weekly for 12 weeks.
  Arms: Stretching and Relaxation

SUMMARY:
This study will compare three different exercise programs in older adults who report difficulty walking and will determine if the programs improve walking.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who live in the lower mainland (greater Vancouver) area of British Columbia
* Aged 65 years or older
* Living independently in their own home
* Report mobility limitation, defined as any difficulty walking one-quarter mile (about 2-3 blocks) outside on level ground or climbing one flight of stairs (about 10 steps) without resting because of a health or physical problem

Exclusion Criteria:

* Have a current medical condition for which exercise is contraindicated
* Have participated in an exercise intervention study in the past 6 months
* Do not have adequate cognitive function to provide informed consent and participate fully in the study
* Do not speak and understand English fluently

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
energy cost of walking | 12 weeks
  assessed by oxygen consumption during treadmill and overground walking
fatigue and fatigability | 12 weeks
  assessed by questionnaire, rated perceived exertion during walking, and decrements in walking performance over time.
daily activity | 12 weeks
  assessed by accelerometry and the Physical Activity Scale for the Elderly
life-space mobility | 12 weeks
  assessed by life-space mobility questionnaire
endurance | 12 weeks
  assessed by the long-distance corridor walk
physical function | 12 weeks
  assessed by standing balance, gait speed, and chair stands

SECONDARY OUTCOMES:
energy cost of walking | 24 weeks
  assessed by oxygen consumption during treadmill and overground walking
fatigue and fatigability | 24 weeks
  assessed by questionnaire, rated perceived exertion during walking, and decrements in walking performance over time
daily activity | 24 weeks
  assessed by accelerometry and the Physical Activity Scale for the Elderly
life-space mobility | 24 weeks
  assessed by the life-space mobility questionnaire
endurance | 24 weeks
  assessed by the long-distance corridor walk
physical function | 24 weeks
  assessed by standing balance, gait speed, and chair stands

CONTACTS AND LOCATIONS:
Overall Officials: Dawn C Mackey, PhD, Principal Investigator — Simon Fraser University; Vancouver Coastal Health Research Institute, Centre for Hip Health and Mobility
Locations (1):
- Centre for Hip Health and Mobility, Vancouver Coastal Health Research Institute, Vancouver, British Columbia, Canada